CLINICAL TRIAL: NCT05031624
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 1 Study of Single Ascending Doses of Subcutaneous CDX-0159 to Assess the Safety, Pharmacokinetics, and Pharmacodynamics in Healthy Subjects
Brief Title: A Phase 1 Study of Subcutaneous CDX-0159 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celldex Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CDX0159-05
Record Dates: First submitted 2021-07-29; First posted 2021-09-02 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Healthy Subjects
Keywords: CDX0159-05
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CDX-0159 (Experimental): Subjects will receive a single dose of CDX-0159
  Interventions: Drug: CDX-0159
- Normal Saline (Placebo Comparator): Subjects will receive a single dose of normal saline
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: CDX-0159 — Single subcutaneous dose of one of four dosages of CDX-0159
  Arms: CDX-0159
Drug: Normal saline — Single subcutaneous dose of normal saline
  Arms: Normal Saline

SUMMARY:
This is a study to determine the safety and pharmacokinetics of CDX-0159 administered subcutaneously in healthy subjects.

DETAILED DESCRIPTION:
CDX-0159 is a humanized monoclonal antibody that binds to a protein called KIT that is expressed on mast cells.

The study will evaluate the safety, pharmacokinetics, and pharmacodynamics of CDX-0159 administered subcutaneously in healthy subjects.

ELIGIBILITY:
Key Inclusion Criteria:

* An informed consent signed and dated by the subject.
* Healthy volunteer aged 18-55.
* In generally good health and without significant medical conditions based on physical exam, ECG, and laboratory test results.
* Body mass index (BMI) ≥ 18.5 kg/m2 to ≤ 35 kg/m2
* No medication other than mild analgesics, vitamins and mineral supplements or, oral contraceptives.
* Both males and females of child bearing potential must agree to use a medically accepted contraceptive regimen during study and up to 150 days afterwards.
* Not a current smoker, vaper, or regular user of any nicotine or cannabinoid containing products
* Willing to follow all study rules

Key Exclusion Criteria:

* Women who are pregnant or nursing
* History of anaphylaxis or systemic reactions to food or other triggers
* Autoimmune disorders requiring more than topical medication
* Vaccination with live vaccines within 4 months prior to screening visit (subjects must agree to avoid live vaccination during the study and 4 months after).
* Positive urine test for alcohol and drugs of abuse.

Other Protocol defined inclusion and exclusion criteria could apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2022-01-14 (Actual); Study Completion 2022-01-14 (Actual)

PRIMARY OUTCOMES:
Safety as assessed by Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Trials | Day 1 to Day 85
  Safety of single, ascending doses of CDX-0159 as determined by percentage of participants with adverse events as assessed by Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Trials

SECONDARY OUTCOMES:
CDX-0159 serum evaluations over time | Day 1 to Day 85
  CDX-0159 serum concentrations will be measured at specified visits
Serum tryptase levels over time | Day 1 to Day 85
  The effect of CDX-0159 on serum tryptase levels
Plasma levels over time | Day 1 to Day 85
  The effect of CDX-0159 on stem cell factor levels
Measurement of Anti-drug Antibody development over time | Day 1 to Day 85
  Patients will be monitored for the development of anti-drug antibodies.

CONTACTS AND LOCATIONS:
Locations (1):
- Celerion, Inc, Lincoln, Nebraska, United States